CLINICAL TRIAL: NCT05727748
Title: Effects of a Multimodal Program With Augmented Reality on Cognition, Functional Fitness and Physical Activity in Older Adults
Brief Title: Effects of an Exercise Program With Augmented Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Évora (Other)
Collaborators: Comprehensive Health Research Center (Other); Foundation for Science and Technology, Portugal (Other)
Responsible Party: Principal Investigator, Soraia Daniela Pires Ferreira, Principal Investigator, University of Évora
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AR_UEvora
Record Dates: First submitted 2023-01-10; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Aging; Older Adults
Keywords: Augmented Reality; Older adults; Exercise; Cogntion
MeSH Terms: conditions — Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: There are three different groups: a) a control group; b) a multimodal training group that combined physical training with cognitive training; c) a multimodal training group with augmented reality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other): The control group continued their daily activities for 12 weeks and did not participate in any new physical activity program during the study.
  Interventions: Other: Control group
- Multimodal training group (Experimental): The session consisted of four stations where participants simultaneously trained physical aspects (cardiorespiratory fitness, strength, balance, and flexibility) and cognitive aspects (reaction time, memory, decision making, semantics, and processing speed).
  Interventions: Other: Multimodal exercise
- Multimodal training group with augmented reality (Experimental): The session consisted of six stations where participants simultaneously trained physical aspects (cardiorespiratory fitness, strength, balance, and flexibility) and cognitive aspects (reaction time, memory, decision making, semantics, and processing speed). Four stations are the same of the previous group and the other 2 stations are with augmented reality. These 2 stations worked the same cognitive and physical components but through the portable exergame platform for the elderly.
  Interventions: Other: Multimodal exercise with augmented reality

INTERVENTIONS:
Other: Multimodal exercise with augmented reality — The intervention program has a duration of 12 weeks with 3 sessions per week of 60 minutes each. The multimodal group with augmented reality was divided into 4 sub-groups. The session consisted of six stations where participants simultaneously trained physical aspects (cardiorespiratory fitness, strength, balance, and flexibility) and cognitive aspects (reaction time, memory, decision making, semantics, and processing speed). Four stations are the same of the previous group and the other 2 stations are with augmented reality. These 2 stations worked the same cognitive and physical components but through the portable exergame platform for the elderly.
  Arms: Multimodal training group with augmented reality
Other: Multimodal exercise — The intervention program has a duration of 12 weeks with 3 sessions per week of 60 minutes each. The multimodal group was divided into 2 sub-groups. The session consisted of four stations where participants simultaneously trained physical aspects (cardiorespiratory fitness, strength, balance, and flexibility) and cognitive aspects (reaction time, memory, decision making, semantics, and processing speed).
  The session consisted of six stations where participants simultaneously trained physical aspects (cardiorespiratory fitness, strength, balance, and flexibility) and cognitive aspects (reaction time, memory, decision making, semantics, and processing speed).
  Arms: Multimodal training group
Other: Control group — The control group continued their daily activities for 12 weeks and did not participate in any new physical activity program during the study.
  Arms: Control group

SUMMARY:
The objectives of the present research is to observe the effects of a multimodal program with augmented reality on cognition, functional fitness, quality of life, and physical activity in older people.

DETAILED DESCRIPTION:
The present investigation lasted 16 weeks. The first two weeks were for familiarization with the tests and initial assessments. This was followed by the 12-week intervention and final assessments (2 weeks).

The intervention program ran for 12 weeks with 3 sessions per week of 60 minutes each. There were three different groups: a) a control group; b) a multimodal training group that combined physical training with cognitive training; c) a multimodal training group with augmented reality.

The control group continued their daily activities for 12 weeks and did not participate in any new physical activity program during the study. In the multimodal training group, the session consisted of four stations where participants simultaneously trained physical aspects (cardiorespiratory fitness, strength, balance, and flexibility) and cognitive aspects (reaction time, memory, decision making, semantics, and processing speed). In the multimodal training session with augmented reality, the session consisted of 6 stations, 4 stations as in the previous group and 2 stations with augmented reality. These 2 stations used the same components but through the portable exergame platform for the elderly.

During the 12 weeks, the intensity and difficulty of each exercise was increased after each session, depending on the evolution of the participants.

When forming the training groups, the participants who were not available during the intervention phase were assigned to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Participants of both genders
* 60 years old or more
* Community-dwelling older adults living independently
* Able to walk autonomously

Exclusion Criteria:

* Having cognitive impairment
* Neurological disorders

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Mini Mental State Examination (MMSE) | 13 weeks
  Evaluates the cognitive state of the participant. The MMSE consists of 6 different domains: orientation, retention, attention and calculation; recall; language, and constructive skills. The maximum score for this test is 30 points. However, the education of the participant education is also taken into account when assigning the score.The scores for determining whether a person has cognitive impairment through the Mini-Mental State Examination (MMSE) are: cut-offs of ≤27 points or persons with >11 years of school education, ≤22 for persons ranging from 1 to 11 years of school education and ≤ 15 points for illiterate persons.
Frontal assessment battery (FAB) | 13 weeks
  Evaluates executive functions, consisting of 6 tests that explore abilities that are related to the frontal lobes. At FAB, the highest score is 18, indicating the best possible performance on the test. The FAB is divided into 6 domains: Conceptualization, Mental Flexibility, Programming, Sensitivity to Interference, Inhibitory Control, and Environmental Autonomy. In each of the subdomains, the score ranges from 0 (worst performance) to 3 (best performance). The subdomains are assessed by short tasks given to the participants.
Deary - Liewald reaction time task | 13 weeks
  Simple and choice reaction time
Trail Making Test | 13 weeks
  Cognitive flexibility and processing speed
Phonemic and semantic verbal fluency test. | 13 weeks
  The test assesses language production, non-motor processing speed, and executive functions.
  In the semantic fluency task, participants had to say as many animals as possible over 60seconds. In the phonemic fluency exercise, participants were asked to list as many words starting with a specific letter as possible. The duration of the exercise was 60seconds. More words correspond to better scores.
Stroop | 13 weeks
  Inhibition and resistance to interference. The stroop test consists of three different tasks, each lasting 45 seconds. In the first task, the participant had to read the words presented, and the words could be red, green, blue, and green. In the second task, participants had to say what color they were seeing (red, green, blue or green). In the last task, participants were presented with several words (red, green, blue, and green) written in different colors and were asked to list the color of ink for each word. The number of correct answers was recorded, with the number of correct answers giving the better score. For the participant to meet the normative data, they should enumerate more than 40 words/colors.

SECONDARY OUTCOMES:
Physical activity | 13 weeks
  Physical activity was measured using accelerometry. Participants wore the accelerometer on their waist for 7 days. Sedentary time, light, moderate, and vigorous physical activity were recorded. At the end, the results reflected the number of minutes per day/week.
Senior Fitness Test - Rikli and Jones | 13 weeks
  This test battery evaluates: cardiorespiratory fitness, strength, endurance, flexibility, agility and balance. It consists of 6 different tests: 30-second chair stand (lower limb strength), arm curl (upper limb strength), chair sit and reach (lower limb flexibility), back scratch (upper limb flexibility), 6-minute walk (cardiorespiratory fitness), 8-foot up-ang-go (agility). For each of the tests there are normative values depending on age and gender.
Body Composition | 13 weeks
  Body composition analyzer - Tanita. Tanita works with an electrical bioimpedance analysis that allows to determine body water, visceral fat, fat mass, lean mass, weight, body mass index, bone mass and muscle mass. This device generates a report that indicates whether the patient is in the healthy range or not.
EQ-5D | 13 weeks
  The 5D questionnaire is used to assess quality of life. It consists of 5 dimensions, mobility, self-care, daily activities, pain, and anxiety/depression. For each dimension, there are 5 response options with a score ranging from 1 (no problem at all) to 5 (unable to do anything).
SF-36 | 13 weeks
  The SF -36 questionnaire is used to assess the participant's health status of participants. It consists of 36 items that assess physical functioning, physical performance, physical pain, emotional functioning, vitality, mental health, social functioning, and general health. The higher the score, the better the participant's health.
Geriatric depression scale | 13 weeks
  The depression scale developed by Yesavage has been used to screen for depression. This scale assesses cognitive and behavioral aspects usually involved in depression in the elderly. We used the short version of the scale with 15 questions in which the responses are dichotomous. One point is assigned for responses indicating depression. Scores between 0 and 5 mean that there is no depression; between 6 and 10 mean that there is mild depression, and 11 and 15 mean that the person has severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Soraia Daniela Pires Ferreira, Leiria, Portugal